CLINICAL TRIAL: NCT06450340
Title: Effects of Tai Chi on Health Fitness and Quality of Life in Youngsters with Visual Impairments: a Randomized Controlled Trial
Brief Title: A Trial of Tai Chi Intervention for Youngsters with Visual Impairments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yanyun Zhang (Other)
Responsible Party: Sponsor-Investigator, Yanyun Zhang, Primary rehabilitation therapist, Guangzhou University of Chinese Medicine
Organization: Guangzhou University of Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PJ-XS-20240422-003
Record Dates: First submitted 2024-06-01; First posted 2024-06-10 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Visual Impairment and Blindness (Excl Colour Blindness)
Keywords: Tai Chi; physical fitness; sleep quality; quality of life
MeSH Terms: conditions — Vision Disorders; Blindness; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tai Chi exercise group (Experimental): Sessions lasted 60 minutes each and took place three times a week for 12 weeks for Tai Chi exercise group.
  Interventions: Behavioral: Moderate-intensity aerobic exercise refers to rhythmic and long-lasting exercise with increased heart rate, slight sweating and slight wheezing.
- Jogging group (Other): Sessions lasted 60 minutes each and took place three times a week for 12 weeks for Jogging group.
  Interventions: Behavioral: Moderate-intensity aerobic exercise refers to rhythmic and long-lasting exercise with increased heart rate, slight sweating and slight wheezing.

INTERVENTIONS:
Behavioral: Moderate-intensity aerobic exercise refers to rhythmic and long-lasting exercise with increased heart rate, slight sweating and slight wheezing. — Sessions lasted 60 minutes each and took place three times a week for 12 weeks for each of the study groups.

SUMMARY:
Investigators conducted a single-blind, randomized trial of Taijiquan exercise as compared with a control intervention consisting of wellness education and jogging for youngsters with visual impairments. Sessions lasted 60 minutes each and took place three times a week for 12 weeks for each of the study groups. The primary end point was a change in the Brockport Physical Fitness Test (BPFT) at the end of 12 weeks. Secondary end points included summary scores of the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) and Pittsburgh Sleep Quality Index (PSQI)at the end of 12 weeks.

DETAILED DESCRIPTION:
* Brockport Physical Fitness Test (BPFT) for youngsters with visual impairments, including 20-meter lap scores, Body mass index (BMI), Dominant Grip Strength, Curl-Up, Trunk lift, Back-Saver Sit-and-Reach and Shoulder Stretch.
* Basic information about visually impaired youth, including age, gender, height, weight.
* summary scores of the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36)
* summary scores of of the Medical Outcomes Study Pittsburgh Sleep Quality Index (PSQI)

ELIGIBILITY:
Inclusion Criteria:

* The age ranges from 10 to 17 years old, regardless of sex.
* had no previous experience as an athlete.
* could follow simple instructions.
* could walk without assistance.
* could maintain a regular lifestyle during the experiment.
* provided informed consent.

Exclusion Criteria:

* The exclusion criterion applied to those who suffered any severe illness or ailment which hinders mobility.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-08 (Actual)

PRIMARY OUTCOMES:
Brockport Physical Fitness Test (BPFT) | One measurement was made from the day of random grouping, and another measurement was made within one week after 12 weeks of exercise intervention.
  BPFT is a physical fitness test for youngsters with disabilities, including a section for youngsters with visual impairments.

SECONDARY OUTCOMES:
36-Item Short-Form Health Survey | One measurement was made from the day of random grouping, and another measurement was made within one week after 12 weeks of exercise intervention.
  Investigators use 36-Item Short-Form Health Survey to test the quality of life of youngsters with visual impairments. The SF-36 is scored on a scale of 0-100, with higher scores indicating better health.
Pittsburgh Sleep Quality Index (PSQI) | One measurement was made from the day of random grouping, and another measurement was made within one week after 12 weeks of exercise intervention.
  Investigators use Pittsburgh Sleep Quality Index (PSQI) to test the sleep quality of youngsters with visual impairments. The total score of the Pittsburgh Sleep Quality Index ranges from 0 to 21, with higher scores indicating worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zheng, Master, Study Director — Master Instructor
Locations (1):
- Guangzhou School For The Visually Impaired, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No